CLINICAL TRIAL: NCT06440720
Title: COMPARATIVE EFFECTS OF ELONGATION LONGITUDINAUX AVEC DECOAPTION OSTEO ARTICULAIRE VERSUS UPPER THORACIC MOBILIZATION AND MOBILITY EXERCISE FOR THE TREATMENT OF FORWARD HEAD POSTURES
Brief Title: COMPARATIVE EFFECTS OF ELDOA VERSES UPPER THORACIC MOBILIZATION AND MOBILITY EXERCISE FOR THE TREATMENT OF FHP
Acronym: ELDOA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Faiza Khalid, FAIZA KHALID, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUF/DR/SA/MSPP/2024/380
Record Dates: First submitted 2024-05-23; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Postural, Thoracic Kyphosis; Postural; Defect
Keywords: Thoracic Mobilization; ELDOA; Mobility Exercise; Posture correction

STUDY DESIGN:
Intervention Model Description: Study Design: Parallel Two-Group Randomized Controlled Trial
  Objective:
  To compare the effectiveness of the Elongation Longitudinaux Avec Decoaptation Osteo Articulaire (ELDOA) method versus upper thoracic mobilization and mobility exercises in treating forward head posture (FHP).
  Participants:
  Total sample size: 36 (18 in each group) Inclusion: Males and females, ages 20-40 years Exclusion: History of neck surgery, severe neck trauma
  Randomization:
  Participants will be randomly assigned to either the ELDOA group or the upper thoracic mobilization group using a computer-generated sequence.
  Interventions:
  Group A (ELDOA): Specific ELDOA exercises for FHP Group B (Upper Thoracic Mobilization): Exercises targeting thoracic mobility and FHP
  Outcome Measures:
  Primary outcomes: Numeric Pain Rating Scale (NPRS), goniometer measurements, Neck Disability Index (NDI), Web Plot Digitizer (WPD) Software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive ELDOA exercises. At first hot pack will applied for 7-8 minutes after that participants will explain specific body movements. Four ELDOA positions will once shown to the participants then ask them to maintain that positions. Once they make these positions stop watch will be set for one minute for each position. these positions will apply for three times per week for four weeks.
  Interventions: Other: ELDOA ,UPPER THORACIC MOBILIZATION AND MOBILITY EXERCISE
- Group-B (Experimental): Group B will receive the UPPER THORACIC MOBILIZATION AND MOBILITY exercise. At first, a hot pack will be applied for 7-8 minutes after that participants will be in a prone position and the physiotherapist will stand toward the side where mobilization will be applied and the index and middle finger of the left hand of the physiotherapist will be placed on the vertebral transverse processes of the participants to the caudal side. The lateral side of the palm of the right hand will be placed over the left-hand index and middle finger and then thoracic mobilization after that mobility exercise will be performed.
  Interventions: Other: ELDOA ,UPPER THORACIC MOBILIZATION AND MOBILITY EXERCISE

INTERVENTIONS:
Other: ELDOA ,UPPER THORACIC MOBILIZATION AND MOBILITY EXERCISE — Already mentioned

SUMMARY:
This study will compare the effectiveness of the Elongation Longitudinaux Avec Decoaptation Osteo Articulaire (ELDOA) method and upper thoracic mobilization and mobility exercises in correcting forward head posture (FHP). This study aims to evaluate the effectiveness of these methods in reducing forward head posture. The total sample size will be 36, with each group consisting of 18 participants. This study will be a randomized clinical trial. Participants who meet the inclusion criteria will be selected through screening and then assessed for outcomes using NPRS, a goniometer, the Neck Disability Index (NDI), and Web Plot Digitizer (WPD) Software. Statistical analysis will be conducted using SPSS version 27.

DETAILED DESCRIPTION:
Study Title Comparative Effectiveness of the ELDOA Method and Upper Thoracic Mobilization and Mobility Exercises in Correcting Forward Head Posture: A Randomized Clinical Trial

Introduction Forward Head Posture (FHP) is a common postural deformity characterized by an anterior positioning of the head relative to the vertical axis of the body. This condition can lead to various musculoskeletal issues, including neck pain, reduced range of motion, and increased disability. The Elongation Longitudinaux Avec Decoaptation Osteo Articulaire (ELDOA) method and upper thoracic mobilization and mobility exercises are two interventions aimed at correcting FHP. This study aims to compare the effectiveness of these two methods in reducing FHP and associated symptoms.

Objectives The primary objective of this study is to evaluate and compare the effectiveness of the ELDOA method and upper thoracic mobilization and mobility exercises in reducing FHP. Secondary objectives include assessing improvements in pain levels, neck disability, and range of motion.

Study Design This study is a randomized clinical trial.

Participants A total of 36 participants will be recruited and randomly assigned to one of two intervention groups, each consisting of 18 participants.

Inclusion Criteria

* Adults aged 20-40 years
* Diagnosed with forward head posture
* Able to provide informed consent
* No history of recent neck or upper thoracic surgery

Exclusion Criteria

* Severe musculoskeletal or neurological disorders
* Recent injury to the neck or upper back
* Pregnant or breastfeeding women

Interventions Group A (ELDOA Method): Participants will undergo the ELDOA method, which involves specific postural exercises designed to create fascial tension and decompress the spine.

Group B (Upper Thoracic Mobilization and Mobility Exercises)**: Participants will receive upper thoracic mobilization techniques combined with mobility exercises aimed at improving posture and reducing FHP.

Outcome Measures

1. Numerical Pain Rating Scale (NPRS): To assess the intensity of pain experienced by participants.
2. Goniometer: To measure the range of motion of the cervical spine.
3. Neck Disability Index (NDI): To evaluate the level of disability associated with neck pain.
4. Web Plot Digitizer (WPD) Software : To analyze and quantify postural changes from photographic data.

Procedure

1. Screening and Baseline Assessment: Participants will be screened for eligibility and baseline measurements will be taken using NPRS, a goniometer, NDI, and WPD.
2. Randomization: Eligible participants will be randomly assigned to either the ELDOA group or the upper thoracic mobilization and mobility exercises group.
3. Intervention Period: Both groups will participate in their respective interventions over a period of 8 weeks, with sessions conducted twice a week.
4. Follow-Up Assessments : Outcomes will be reassessed at the end of the intervention period and compared to baseline values.

Statistical Analysis Data will be analyzed using SPSS version 27. Descriptive statistics will be used to summarize baseline characteristics. Paired t-tests or Wilcoxon signed-rank tests will be used to compare pre- and post-intervention outcomes within groups. Independent t-tests or Mann-Whitney U tests will be employed to compare outcomes between the two groups. A significance level of p < 0.05 will be considered statistically significant.

Expected Outcomes It is hypothesized that both interventions will result in significant improvements in FHP, pain reduction, and decreased neck disability. However, the study aims to determine if one method is superior in achieving these outcomes.

Ethical Considerations This study will adhere to ethical guidelines for clinical research. Informed consent will be obtained from all participants, and the study protocol will be reviewed and approved by an appropriate ethics committee.

Conclusion This randomized clinical trial will provide valuable insights into the comparative effectiveness of the ELDOA method and upper thoracic mobilization and mobility exercises in correcting forward head posture. The findings could inform clinical practice and guide the development of targeted interventions for FHP.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females.
* Age between 20 to 40 years.
* Patients having complain of neck pain
* Patients having forward head posture
* Patients having limited Cervical range of motion
* Patients having Craniovertebral angle CVA less than 50.
* Pain more than 3 on NPRS scale with FHP

Exclusion Criteria:

* History of whiplash injury within 3 months of examination.
* History of tumor
* History of surgery of cervical or thoracic spine.
* Positive neurological signs
* Congenital deformity
* Patients having pathology and infection in spine.
* Patients having severe osteoporosis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral angle | 5 Minutes
  The primary outcome measure was the CVA, which was calculated using each participant's profile photo. The self-balanced posture assessment method was used to force the participants to maintain their typical head posture. By drawing a vertical line from Targus to the seventh cervical vertebrae and a horizontal line across them, the angle between them may be calculated to determine the CVA angle. The CVA measurement was shown to have excellent reliability in a prior research.

SECONDARY OUTCOMES:
Cervical ranges of motion | 20 Minutes
  Cervical ranges of motion ( CROM) cervical flexion, extension, right Side bending, left Side bending, right rotation and left rotation were measured using goniometer
Numeric Pain Rating Scale | 5 Minutes
  The NPRS scale, which has good reliability and validity in prior research, was utilized to measure the degree of present pain. 0: No pain
  1 - 3: Mild pain 4 - 6: Moderate pain 7 - 10: Severe pain
Neck disability Index | 10 minutes
  The cervical spine's disability index was assessed using the NDI. It consists of 10 items, each scored on a 0 to 5 scale, with the total score ranging from 0 to 50. The NDI score can be expressed as a percentage by multiplying the raw score by 2. The interpretation of the NDI score is typically as follows:
  0 - 4 (0% - 8%): No disability 5 - 14 (10% - 28%): Mild disability 15 - 24 (30% - 48%): Moderate disability 25 - 34 (50% - 68%): Severe disability 35 - 50 (70% - 100%): Complete disability

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Khalid, MSPT, Principal Investigator — The University of Faisalabad
Locations (1):
- Govt Teaching Hospital GM Abad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kripa S KH. Identifying relations between posture and pain in lower back pain patients: a narrative review. Bulletin of Faculty of Physical Therapy.
- [Background] Waqar S, Faculty of Rehabilitation & Allied Health Sciences RIU, Islamabad. Pakistan, Khalid M, Faculty of Rehabilitation & Allied Health Sciences RIU, Islamabad. Pakistan, Khalid N, Islamabad Physiotherapy & Rehabilitation Centre BT. EFFECTIVENESS OF ELONGATION LONGITUDINAUX AVEC DECOAPTION OSTEOARTICULAIRE IN CORRECTING FORWARD HEAD POSTURE. The Rehabilitation Journal. 2022;volume no.6.
- [Background] Cho J, Lee E, Lee S. Upper thoracic spine mobilization and mobility exercise versus upper cervical spine mobilization and stabilization exercise in individuals with forward head posture: a randomized clinical trial. BMC Musculoskelet Disord. 2017 Dec 12;18(1):525. doi: 10.1186/s12891-017-1889-2. PMID 29233164
- [Result] Weon JH, Oh JS, Cynn HS, Kim YW, Kwon OY, Yi CH. Influence of forward head posture on scapular upward rotators during isometric shoulder flexion. J Bodyw Mov Ther. 2010 Oct;14(4):367-74. doi: 10.1016/j.jbmt.2009.06.006. Epub 2009 Jul 22. PMID 20850044
- [Result] Farooq M, Bashir MS, Arif A, Kashif M, Manzoor N, Abid F. Effects of elongation longitudinaux avec decoaption osteo-articulaire and post-facilitation stretching technique on pain and functional disability in mobile users with text neck syndrome during COVID-19 pandemic: A randomized controlled trial. Medicine (Baltimore). 2023 Mar 24;102(12):e33073. doi: 10.1097/MD.0000000000033073. PMID 36961169